CLINICAL TRIAL: NCT05251103
Title: Time-restricted Feeding Increases Fat Oxidation Rate But Not Affect Postprandial Lipemia: a Crossover Trial
Brief Title: The Effect of Different Methods for Modulating Postprandial Fat Oxidation on Postprandial Lipemia the Next Day
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan Sport University (Other)
Responsible Party: Principal Investigator, Chih-Hui Chiu, Associate Professor, National Taiwan Sport University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 110-10
Record Dates: First submitted 2022-02-02; First posted 2022-02-22 (Actual); Last update posted 2022-02-22 (Actual); Status verified 2022-02

CONDITIONS: Time-restricted Feeding; Postprandial Lipemia
Keywords: intermittent fasting
MeSH Terms: conditions — Intermittent Fasting

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- time-restricted feeding trial (Experimental): The participants were divided into the time-restricted feeding trial for 5 days
  Interventions: Other: time-restricted feeding trial
- control trial (Experimental): The participants in the control trial did not practice intermittent fasting methods
  Interventions: Other: time-restricted feeding trial

INTERVENTIONS:
Other: time-restricted feeding trial — The 5-day time-restricted feeding trial and the control trial. The meals of the time-restricted feeding trial were provided at 12:00, 16:00, and 20:00.

SUMMARY:
Background: Studies have revealed that time-restricted feeding affects the fat oxidation rate; however, its effects on the fat oxidation rate and hyperlipidemia following high-fat meals are unclear. This study investigated the effects of 5-day time-restricted feeding on the fat oxidation rate and postprandial lipemia following high fat meals. Methods: In this random crossover experimental study, eight healthy male adults were included each in the 5-day time-restricted feeding trial and the control trial. The meals of the time-restricted feeding trial were provided at 12:00, 16:00, and 20:00. The meals of the control trial were provided at 08:00, 14:00, and 20:00. The contents of the meals of both trials were the same, and the calories of the meals met the 24-hour energy requirement of the participants. After 5 days of the intervention, the participants consumed high-fat meals on the sixth day, and their physiological changes were determined.

DETAILED DESCRIPTION:
The experiment was conducted over 6 days. On the first day, the participants arrived at the laboratory at 08:00 and quietly rested for 20 minutes in the supine position; gas analyzers were used to record their energy consumption. Subsequently, the participants were randomly allocated to the time-restricted feeding trial or the control trial. The meals of the time-restricted feeding trial were provided at 12:00, 16:00, and 20:00, and the participants were required to consume all the food during this time. The meals of the control trial were provided at 08:00, 14:00, and 20:00, but the consumption time was not limited. In addition to regular meals, a snack with approximately 200 calories was provided to the participants for consumption. The participants in the time-restricted feeding trial were only allowed to consume the snack from 12:00 to 20:00, whereas no restrictions were imposed on the control trial for snack consumption. The meals of the participants were provided by dieticians. Based on the results of the pretest, the calories of each meal met the daily energy requirement of the participants. The macronutrient consumption for TRF and CON were listed in table 1.

After experiment completion on the fifth day, the participants returned to the laboratory on the eighth day from 08:00 to 09:00. They rested for 10 minutes in the supine position, and gas analyzers were used to collect the gas data of the participants for 20 minutes. Next, a catheter was inserted into the forearm of each participant to collect fasting blood samples. After blood sample collection, the participants were provided with a specific high-fat meal. The participants rested quietly in the laboratory for 4 hours, and their blood lipid changes during this period were observed.

ELIGIBILITY:
Inclusion Criteria:

* All the participants had not undergone physical training;
* they did not exercise regularly;
* and they did not have any diseases that would prevent them from performing exercises, such as high blood pressure, hyperlipidemia, heart disease, joint disease, and osteoporosis.

Exclusion Criteria:

* Undergone physical training;
* Exercise regularly;
* Have any diseases that would prevent them from performing exercises, such as high blood pressure, hyperlipidemia, heart disease, joint disease, and osteoporosis.

Min Age: 20 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2021-06-04 (Actual); Primary Completion 2022-02-03 (Actual); Study Completion 2022-02-03 (Actual)

PRIMARY OUTCOMES:
postprandial triglycerides concentrations | on the 6th day
  postprandial triglycerides concentrations (mmol/L)
postprandial glucose concentrations | on the 6th day
  postprandial glucose concentrations (mmol/L)
postprandial insulin concentrations | on the 6th day
  postprandial insulin concentrations (pmol/L)
postprandial free fatty acid concentrations | on the 6th day
  postprandial FFA concentrations (mmol/L)
postprandial glycerol concentrations | on the 6th day
  postprandial glycerol concentrations (umol/L)

SECONDARY OUTCOMES:
fat oxidation | on the 6th day
  fasting fat oxidation rate (g/min-1)

CONTACTS AND LOCATIONS:
Overall Officials: ChihHui Chiu, PhD, Study Chair — National Taiwan University of Sport
Locations (1):
- National Taiwan University of Sport, Taichung, Taiwan

DOCUMENTS (1):
  • Study Protocol (2022-02-02): https://cdn.clinicaltrials.gov/large-docs/03/NCT05251103/Prot_000.pdf